CLINICAL TRIAL: NCT02856581
Title: Reducing Surgical Complications in Newly Diagnosed Lung Cancer Patients Who Smoke Cigarettes
Brief Title: Management of Tobacco Treatment Intervention in Reducing Surgical Complications in Patients With Newly Diagnosed Lung Cancer Who Smoke Cigarettes
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: A211401; NCI-2016-00438 (Registry Identifier: NCI Clinical Trial Reporting Program)
Record Dates: First submitted 2016-08-01; First posted 2016-08-05 (Estimated); Results first posted 2022-06-24 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-06

CONDITIONS: Lung Carcinoma
MeSH Terms: conditions — Lung Neoplasms | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention group (varenicline and behavioral intervention) (Experimental): Patients receive varenicline PO QD on days 1-3 and BID on days 4-84 for 12 weeks in the absence of disease progression or unacceptable toxicity. Patients also complete behavioral intervention consisting of no smoking message from surgical team member and how to use NCI quitline at surgical consult.
  Interventions: Drug: Varenicline; Other: Tobacco Cessation Counseling
- Control group (placebo and behavioral intervention) (Placebo Comparator): Patients receive placebo PO QD on days 1-3 and BID on days 4-84 for 12 weeks in the absence of disease progression or unacceptable toxicity. Patients also complete behavioral intervention consisting of no smoking message from surgical team member and how to use NCI quitline at surgical consult.
  Interventions: Drug: Placebo; Other: Tobacco Cessation Counseling

INTERVENTIONS:
Drug: Varenicline — Given PO
  Arms: Intervention group (varenicline and behavioral intervention)
Drug: Placebo — Given PO
  Arms: Control group (placebo and behavioral intervention)
Other: Tobacco Cessation Counseling — Complete counseling session

SUMMARY:
This randomized phase III trial studies how well management of a tobacco treatment intervention works in reducing surgical complications in patients with newly diagnosed lung cancer who smoke cigarettes. Management of a tobacco treatment intervention compares varenicline (a drug that reduces the craving and withdrawal symptoms that occur with abstinence from nicotine) and behavioral interventions (consisting of a brief clinician-delivered intervention and tobacco quitline [tobacco cessation service available through a toll-free telephone number] follow-up) with placebo (a pill with no active medication) along with similar behavioral interventions. It is not yet known whether management of a tobacco treatment intervention is more effective in reducing surgical complications than placebo.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if varenicline plus a behavioral intervention consisting of a brief clinician-delivered intervention and tobacco quitline follow-up, decreases postsurgical complications through 24 weeks after surgery when compared to placebo plus the behavioral intervention in lung cancer patients who undergo surgery and are motivated to stop smoking.

SECONDARY OBJECTIVES:

I. To compare changes from baseline to 12 and 24 weeks after surgery in the patient quality of life (Linear Analogue Self-Assessment [LASA]-12) domains between the intervention (varenicline) and control group (placebo).

II. To compare changes from baseline to 6, 12 and 24 weeks after surgery in the patient quality of life related domains (LASA) for the Patient Health Questionnaire (PHQ)-9 and Smoking Self Efficacy Questionnaire (SEQ)12 between the intervention and control groups.

III. To compare the proportion of patients 12 weeks and 24 weeks after surgery who endorse ("Was It Worth It") each treatment (intervention versus [vs] control groups).

IV. To compare post-operative care (as measured by length of hospital and high dependency unit stay) between the intervention and control groups.

V. To compare treatment adherence between the intervention and control groups. VI. To compare rates of smoking abstinence between the intervention and control groups as a covariate of the primary outcome only.

ELIGIBILITY:
* Eligible patients will have a new diagnosis of lung cancer and have sought a surgical consult relating to this diagnosis
* Surgery must be scheduled no sooner than 10 days after randomization and no more than twelve weeks after randomization
* Have smoked daily or nearly every day in the previous 6 months up to the date of surgical consult AND have smoked at least one puff in the previous 7 days
* Motivated to stop smoking, as indicated by a score of 6 or above on the Contemplation Ladder
* Within the 30 days before registration, no use of: 1) any pharmacologic treatment for smoking cessation, including bupropion or nicotine replacement therapy; 2) any nicotine delivery system (i.e., e-cigarettes and vape products); or 3) be enrolled in any formal behavioral treatment program for tobacco dependence as determined by patient report
* No allergies to and not currently using varenicline
* No suicidal thoughts as indicated by a positive (1+) response to the PHQ9
* No active untreated clinically significant psychiatric condition (psychosis, bipolar disorder, or depression)
* Negative pregnancy test (serum or urine) done =< 7 days prior to registration, for women of childbearing potential only

  * A female of childbearing potential is a sexually mature female who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months)
* No unstable angina, myocardial infarction, or coronary angioplasty within the past 3 months or an untreated cardiac dysrhythmia
* No history of seizures
* No unstable neurologic, hepatic, renal, cardiovascular, lymphatic, or metabolic disease
* Not currently on renal dialysis or has a history of significant renal impairment
* No recent history (=< 90 days) of substance abuse (outside of tobacco) defined by National Institute on Alcohol Abuse and Alcoholism (NIAAA) as:

  * If male, drinking > 14 alcoholic beverages per week for past 1 month
  * If female, drinking > 7 alcoholic beverages per week for past 1 month
  * Use of cocaine, heroin, club drugs (i.e., 3,4-methylenedioxymethamphetamine (MDMA)/"ecstasy"), methamphetamine, or hallucinogens (e.g., lysergic acid diethylamide [LSD]) at any time during the past 1 month
  * Use of marijuana on a weekly basis for the past 1 month
* Patients must be able to complete study questionnaires in English
* No other household member or relative participating in the study
* No known history of any condition or factor judged by the investigator to preclude participation in the study or which might hinder study adherence
* Calculated creatinine clearance >= 30 mL/min * For females, use 85% of calculated creatinine clearance (CrCl) value

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-09-29 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2022-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ivana Croghan, PhD, Study Chair — Mayo
Locations (374):
- United States (374):
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Kingman Regional Medical Center, Kingman, Arizona
  - Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - PCR Oncology, Arroyo Grande, California
  - Veterans Affairs Loma Linda Healthcare System, Loma Linda, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - Saint Helena Hospital, St. Helena, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - Cancer Center of Colorado at Sloan's Lake, Denver, Colorado
  - National Jewish Health-Main Campus, Denver, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western Surgical Care, Denver, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Good Samaritan Medical Center, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - McKee Medical Center, Loveland, Colorado
  - National Jewish Health-Northern Hematology Oncology, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Middlesex Hospital, Middletown, Connecticut
  - Veterans Affairs Connecticut Healthcare System-West Haven Campus, West Haven, Connecticut
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Memorial Hospital West, Pembroke Pines, Florida
  - Indian River Medical Center, Vero Beach, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Summit Cancer Care-Candler, Savannah, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Alphonsus Medical Center-Nampa, Nampa, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Northwest Community Hospital, Arlington Heights, Illinois
  - Rush - Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Marjorie Weinberg Cancer Center at Loyola-Gottlieb, Melrose Park, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Cancer Care Specialists of Illinois-Swansea, Swansea, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Deaconess Clinic Downtown, Evansville, Indiana
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - Parkview Regional Medical Center, Fort Wayne, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - Franciscan Health Mooresville, Mooresville, Indiana
  - Chancellor Center for Oncology, Newburgh, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Baptist Health Corbin, Corbin, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - Baptist Health Madisonville/Merle Mahr Cancer Center, Madisonville, Kentucky
  - Baptist Health Paducah, Paducah, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Medical Center of Baton Rouge, Baton Rouge, Louisiana
  - Ochsner High Grove, Baton Rouge, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - UM Upper Chesapeake Medical Center, Bel Air, Maryland
  - Mercy Medical Center, Springfield, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - IHA Hematology Oncology Consultants-Brighton, Brighton, Michigan
  - Saint Joseph Mercy Brighton, Brighton, Michigan
  - IHA Hematology Oncology Consultants-Canton, Canton, Michigan
  - Saint Joseph Mercy Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - IHA Hematology Oncology Consultants-Chelsea, Chelsea, Michigan
  - Saint Joseph Mercy Chelsea, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Beaumont Hospital - Dearborn, Dearborn, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Great Lakes Cancer Management Specialists-Doctors Park, East China Township, Michigan
  - Genesee Cancer and Blood Disease Treatment Center, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Academic Hematology Oncology Specialists, Grosse Pointe Woods, Michigan
  - Great Lakes Cancer Management Specialists-Van Elslander Cancer Center, Grosse Pointe Woods, Michigan
  - Michigan Breast Specialists-Grosse Pointe Woods, Grosse Pointe Woods, Michigan
  - Allegiance Health, Jackson, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Medical Campus, Macomb, Michigan
  - Michigan Breast Specialists-Macomb Township, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - UP Health System Hematology Oncology Marquette, Marquette, Michigan
  - UP Health System Marquette, Marquette, Michigan
  - 21st Century Oncology-Pontiac, Pontiac, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Huron Medical Center PC, Port Huron, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Great Lakes Cancer Management Specialists-Rochester Hills, Rochester Hills, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - Ascension Saint Joseph Hospital, Tawas City, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Professional Building, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Michigan Breast Specialists-Warren, Warren, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - IHA Hematology Oncology Consultants-Ann Arbor, Ypsilanti, Michigan
  - Mayo Clinic Health Systems-Mankato, Mankato, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Saint Cloud Hospital, Saint Cloud, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Golden Triangle, Columbus, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Singing River Hospital, Pascagoula, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Hospital, Missoula, Montana
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - 21st Century Oncology-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Las Vegas Urology - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pebble, Henderson, Nevada
  - Urology Specialists of Nevada - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pecos, Las Vegas, Nevada
  - Desert West Surgery, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - OptumCare Cancer Care at Oakey, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Urology Specialists of Nevada - Central, Las Vegas, Nevada
  - 21st Century Oncology, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Las Vegas Prostate Cancer Center, Las Vegas, Nevada
  - Las Vegas Urology - Sunset, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - 21st Century Oncology-Vegas Tenaya, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Las Vegas Urology - Cathedral Rock, Las Vegas, Nevada
  - Las Vegas Urology - Smoke Ranch, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Urology Specialists of Nevada - Northwest, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - 21st Century Oncology-Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Urology Specialists of Nevada - Southwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Ocean Medical Center, Brick, New Jersey
  - Hunterdon Medical Center, Flemington, New Jersey
  - The Cancer Institute of New Jersey Hamilton, Hamilton, New Jersey
  - Bayshore Community Hospital, Holmdel, New Jersey
  - Southern Ocean County Medical Center, Manahawkin, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Riverview Medical Center/Booker Cancer Center, Red Bank, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - Glens Falls Hospital, Glens Falls, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Vassar Brothers Medical Center, Poughkeepsie, New York
  - University of Rochester, Rochester, New York
  - East Carolina University, Greenville, North Carolina
  - Alliance Cancer Center, Alliance, Ohio
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Saint Elizabeth Boardman Hospital, Boardman, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC-Miami Valley Hospital North, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - First Dayton Cancer Care, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Dayton Physicians LLC-Upper Valley, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Joseph Warren Hospital, Warren, Ohio
  - Saint Elizabeth Youngstown Hospital, Youngstown, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Alphonsus Medical Center-Baker City, Baker City, Oregon
  - Saint Alphonsus Medical Center-Ontario, Ontario, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Medical Oncology-Selinsgrove, Selinsgrove, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Ralph H Johnson VA Medical Center, Charleston, South Carolina
  - Prisma Health Cancer Institute - Laurens, Clinton, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Spartanburg, South Carolina
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Baptist Memorial Hospital for Women, Memphis, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - UTMB Cancer Center at Victory Lakes, League City, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Riverton Hospital, Riverton, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Medical Center Regional Cancer Center, St. George, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Sentara Martha Jefferson Hospital, Charlottesville, Virginia
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Augusta Health Center for Cancer and Blood Disorders, Fishersville, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Virginia Mason Bainbridge Island Medical Center, Bainbridge Island, Washington
  - Overlake Hospital Medical Center, Bellevue, Washington
  - Virginia Mason Federal Way Medical Center, Federal Way, Washington
  - Tacoma/Valley Radiation Oncology Centers-Gig Harbor, Gig Harbor, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Northwest Cancer Clinic, Kennewick, Washington
  - Virginia Mason Lynnwood Medical Center, Lynnwood, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - Peninsula Cancer Center, Poulsbo, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Tacoma/Valley Radiation Oncology Centers-Puyallup, Puyallup, Washington
  - Valley Medical Center, Renton, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Rockwood Cancer Treatment Center-DHEC-Downtown, Spokane, Washington
  - Rockwood North Cancer Treatment Center, Spokane, Washington
  - Rockwood Clinic Cancer Treatment Center-Valley, Spokane Valley, Washington
  - Tacoma/Valley Radiation Oncology Centers-Jackson Hall, Tacoma, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Tacoma/Valley Radiation Oncology Centers-Saint Joe's, Tacoma, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Group (Varenicline and Behavioral Intervention): Patients receive varenicline PO QD on days 1-3 and BID on days 4-84 for 12 weeks in the absence of disease progression or unacceptable toxicity. Patients also complete behavioral intervention consisting of no smoking message from surgical team member and how to use NCI quitline at surgical consult.> > Varenicline: Given PO>
  > Tobacco Cessation Counseling: Complete counseling session
- Control Group (Placebo and Behavioral Intervention): Patients receive placebo PO QD on days 1-3 and BID on days 4-84 for 12 weeks in the absence of disease progression or unacceptable toxicity. Patients also complete behavioral intervention consisting of no smoking message from surgical team member and how to use NCI quitline at surgical consult.> > Placebo: Given PO>
  > Tobacco Cessation Counseling: Complete counseling session
Period: Overall Study
Arm/Group | Intervention Group (Varenicline and Behavioral Intervention) | Control Group (Placebo and Behavioral Intervention)
Started | 12 | 11
Completed | 12 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group (Varenicline and Behavioral Intervention) | Control Group (Placebo and Behavioral Intervention) | Total
Number analyzed (Participants) | 12 | 11 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (7.3) | 63.9 (7.4) | 65.1 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 8
  Male | 10 | 5 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 8 | 8 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 11 | 23

OUTCOME MEASURES:

1. Primary Outcome: Mortality
Description: Number of patients that died within 30 days of surgery
Time Frame: Up to 30 days post-surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group (Varenicline and Behavioral Intervention) | Control Group (Placebo and Behavioral Intervention)
Number analyzed (Participants) | 12 | 11
Participants | 0 | 0

2. Primary Outcome: Re-hospitalization
Description: Number of patients re-hospitalized within 30 days of surgery
Time Frame: Up to 30 days post-surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group (Varenicline and Behavioral Intervention) | Control Group (Placebo and Behavioral Intervention)
Number analyzed (Participants) | 12 | 11
Participants | 0 | 0

3. Primary Outcome: Number of Paticipants With Incidence of Pulmonary Complications
Description: Surgical complication incidence rates at 24 weeks after surgery will be compared between the intervention vs. control groups using a Fisher's exact test. Logistic regression models will supplement the univariate analysis, using complication incidence as the dependent variable and will include smoking status at the time of surgery as an independent variable and also adjust for age, gender, Fagerström Test for Nicotine Dependence (FTND), time between randomization and surgery, and presence of adjuvant chemotherapy and/or radiation therapy. We will also explore the collinear relationship between arm and smoking status to see whether they can be included together in the logistic models.
Time Frame: Up to 24 weeks post-surgery
Measure: Count of Participants; unit: Participants
Groups:
- Intervention Group (Varenicline and Behavioral Intervention): Patients receive varenicline PO QD on days 1-3 and BID on days 4-84 for 12 weeks in the absence of disease progression or unacceptable toxicity. Patients also complete behavioral intervention consisting of no smoking message from surgical team member and how to use NCI quitline at surgical consult.
  >
  > Varenicline: Given PO
  >
  > Tobacco Cessation Counseling: Complete counseling session
- Control Group (Placebo and Behavioral Intervention): Patients receive placebo PO QD on days 1-3 and BID on days 4-84 for 12 weeks in the absence of disease progression or unacceptable toxicity. Patients also complete behavioral intervention consisting of no smoking message from surgical team member and how to use NCI quitline at surgical consult.
  >
  > Placebo: Given PO
  >
  > Tobacco Cessation Counseling: Complete counseling session
Arm/Group | Intervention Group (Varenicline and Behavioral Intervention) | Control Group (Placebo and Behavioral Intervention)
Number analyzed (Participants) | 12 | 11
Participants | 0 | 0

4. Primary Outcome: Number of Participants With Incidence of Intensive Care Unit Readmission
Description: Surgical complication incidence rates at 24 weeks after surgery will be compared between the intervention vs. control groups using a Fisher's exact test. Logistic regression models will supplement the univariate analysis, using complication incidence as the dependent variable and will include smoking status at the time of surgery as an independent variable and also adjust for age, gender, FTND, time between randomization and surgery, and presence of adjuvant chemotherapy and/or radiation therapy. A separate logistic model will be created including treatment arm instead of smoking status. We will also explore the collinear relationship between arm and smoking status to see whether they can be included together in the logistic models.
Time Frame: Up to 24 weeks post-surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group (Varenicline and Behavioral Intervention) | Control Group (Placebo and Behavioral Intervention)
Number analyzed (Participants) | 12 | 11
Participants | 0 | 0

5. Primary Outcome: Number of Participants With Incidence of Unspecified Wound Infection
Description: as for outcome 4
Time Frame: Up to 24 weeks post-surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group (Varenicline and Behavioral Intervention) | Control Group (Placebo and Behavioral Intervention)
Number analyzed (Participants) | 12 | 11
Participants | 0 | 0

6. Primary Outcome: Number of Participants With Incidence of Anastomotic Failure
Description: as for outcome 4
Time Frame: Up to 24 weeks post-surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group (Varenicline and Behavioral Intervention) | Control Group (Placebo and Behavioral Intervention)
Number analyzed (Participants) | 12 | 11
Participants | 0 | 0

7. Secondary Outcome: Change in QOL as Measured by the LASA-12, PHQ-9, SEQ-12
Description: Analysis of covariance and linear mixed model repeated measures analysis will be used for each assessment domain (LASA-12, PHQ-9, SEQ12).
Time Frame: Baseline up to 24 weeks after surgery
Reporting Status: Not Posted

8. Secondary Outcome: Change in QOL as Measured by Was It Worth It Assessments
Time Frame: At 12 weeks after surgery
Reporting Status: Not Posted

9. Secondary Outcome: Change in QOL as Measured by Was It Worth It Assessments
Time Frame: At 24 weeks after surgery
Reporting Status: Not Posted

10. Secondary Outcome: Length of Hospital Stay
Description: Logrank testing of Kaplan-Meier estimates will be used for length of hospital stay and supplemented by Cox models to control for concomitant covariates.
Time Frame: The time from surgery until the patient is released from the hospital
Reporting Status: Not Posted

11. Secondary Outcome: Length of High Dependency Unit Stay
Description: Logrank testing of Kaplan-Meier estimates will be used for length of high dependency unit stay and supplemented by Cox models to control for concomitant covariates.
Time Frame: The time from surgery until the patient is released from the hospital
Reporting Status: Not Posted

12. Secondary Outcome: Expanded Complication Rate
Time Frame: Up to 1 year
Reporting Status: Not Posted

13. Secondary Outcome: Treatment Adherence Rates Related to Visits, Medication Compliance, Quitline Usage, and Surgeon Teachable Moment Delivery
Time Frame: Up to 12 weeks
Reporting Status: Not Posted

14. Secondary Outcome: Smoking Abstinence Rates as Measured by Self-report
Time Frame: Up to 12 weeks
Reporting Status: Not Posted

15. Secondary Outcome: Smoking Abstinence Rates as Measured by Salivary Cotinine Testing
Time Frame: Up to 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Intervention Group (Varenicline and Behavioral Intervention) | Control Group (Placebo and Behavioral Intervention)
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/12 | 2/11
Other Adverse Events (participants affected / at risk) | 2/12 | 4/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Group (Varenicline and Behavioral Intervention) (N=12) | Control Group (Placebo and Behavioral Intervention) (N=11)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (2)
Gen disord and admin site conds-Oth spec (General disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Group (Varenicline and Behavioral Intervention) (N=12) | Control Group (Placebo and Behavioral Intervention) (N=11)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Edema face (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (3)
Gen disord and admin site conds-Oth spec (General disorders) | 0 (0) | 1 (1)
Personality change (Psychiatric disorders) | 1 (1) | 0 (0)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-27): https://cdn.clinicaltrials.gov/large-docs/81/NCT02856581/Prot_SAP_000.pdf